CLINICAL TRIAL: NCT00357773
Title: Clinical Efficacy and Safety of T1225 1.5% Eye Drops (3-Day Treatment) Versus Tobramycin 0.3 % Eye Drops (7-Day Treatment) in the Treatment of Purulent Bacterial Conjunctivitis
Brief Title: Efficacy and Safety of T1225 1.5% Versus Tobramycin 0.3 % in the Treatment of Purulent Bacterial Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT1225-PIII-11/03
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2006-07

CONDITIONS: Conjunctivitis, Bacterial
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin (T1225)

SUMMARY:
To demonstrate the efficacy of T1225 1.5% eye drops, in comparison to reference product, for the treatment of purulent bacterial conjunctivitis, and to assess the safety

DETAILED DESCRIPTION:
The aim of the present study was to compare the efficacy and safety of T1225 1.5% eye drops administered BID for 3 days in comparison to reference antibiotic eye drops, tobramycin, for the treatment of purulent bacterial conjunctivitis. The study was conducted as a Phase III, multicentre, international, investigator-masked, randomised, parallel-group, non-inferiority study in newborns, children, and adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >= 1 day old (newborn, infant, child, adult);
* written informed consent by patient or legally acceptable representative;
* purulent bacterial conjunctivitis (unilateral or bilateral) defined as bulbar conjunctival injection (mild, moderate, or severe) AND conjunctival purulent discharge (mild, moderate or severe).

Exclusion Criteria:

* Bacterial conjunctivitis diagnosed >= 7 days ago;
* bacterial infection due to trauma or foreign body;
* dacryocystitis;
* corneal ulceration or keratitis;
* viral ocular infection; closed angle glaucoma;
* acute allergy conjunctivitis;
* clinically significant ocular abnormality;
* organic amblyopia, monophthalmia;
* corrected visual acuity below 20/100;
* contact lens wearer;
* newborn (i.e. 0-2 months old) not born at term (< 37 weeks of amenorrhea);
* ocular surgery, laser in situ keratomileusis (LASIK), laser epithelial keratomileusis (LASEK), or photo-refractive keratectomy (PRK) in last 12 months;
* ocular laser treatment in last 3 months;
* systemic macrolide antibiotics in last month;
* systemic steroids in last 2 weeks or during the study;
* topical ocular macrolide antibiotics and/or topical ocular steroids and/or non-steroidal anti-inflammatory drugs (NSAIDs) in last week;
* topical (ocular, nasal, bronchial etc.) treatments and/or systemic NSAIDs in last day;
* immunosuppressives and/or any systemic antibiotic on D0.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-05; Study Completion 2005-06

PRIMARY OUTCOMES:
Clinical cure in the worse eye on Test of Cure (TOC) visit at Day 9, defined as a score 0 for bulbar conjunctival injection and a score 0 for conjunctival purulent discharge (each graded on 4-point scales)

SECONDARY OUTCOMES:
Clinical cure at Day 3
Microbiological cure at Day 3 and Day 9
Global efficacy.
Tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle COCHEREAU, Professor, Principal Investigator — CHU d'Angers, France